CLINICAL TRIAL: NCT01739582
Title: An Open Label, 6 Month Phase III Extension Study of Enclomiphene Citrate in the Treatment of Men With Secondary Hypogonadism
Brief Title: An Extension Study of Enclomiphene Citrate in the Treatment of Men With Secondary Hypogonadism
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZA-301EXT
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Androxal (Experimental): Androxal (enclomiphene citrate) 12.5 mg, once daily, oral capsule. Subjects will be up-titrated to 25 mg if testosterone levels remain below 450 ng/dL at visit 2.
  Interventions: Drug: Androxal

INTERVENTIONS:
Drug: Androxal
  Other Names: enclomiphene citrate

SUMMARY:
To determine the safety profile of Androxal in men with secondary hypogonadism.

DETAILED DESCRIPTION:
This study is an open-label, multi-center Phase 3 extension study to evaluate the safety on continued treatment with Androxal in subjects who completed either ZA-301 or ZA-302. The study requires 6 study visits (1 for an eye exam) and is approximately 7 months in duration. Subjects will be treated for 26 weeks, starting at a daily dose of 12.5 mg. At Visit 2 (Week 6) subjects who do not achieve morning T values ≥450 ng/dL will be up-titrated to 25 mg. Safety will be assessed by physical and visual acuity exams, slit lamp and fundoscopy, refraction eye exams, clinical laboratory tests and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

• Successful completion of either ZA-301 or ZA-302

Exclusion Criteria:

• Any condition which, in the opinion of the Investigator, would make the Subject an unsuitable candidate for enrollment in the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Testosterone levels | 26 weeks
  Values of total morning testosterone levels at each visit

SECONDARY OUTCOMES:
Follicle Stimulating Hormone and Leutinizing Hormone | 26 weeks
  Values of Follicle Stimulating Hormone (FSH) and Leutinizing Hormone (LH) at each visit
Diabetic Parameters | 26 weeks
  Changes in HbA1c, fasting plasma glucose (FPG), insulin, and homeostasis model assessment-insulin resistance (HOMA-IR) for those subjects with Type II diabetes
Change in weight and body mass index (BMI) | 26 weeks
  Change in weight and BMI

REFERENCES:
- See also: Sponsor corporate web page — http://reprosrx.com